CLINICAL TRIAL: NCT04659083
Title: How NAVA Works in Preterm Infants With Irregular Respiratory Efforts
Status: Completed | Type: Observational
Sponsor: Inha University Hospital (Other)
Collaborators: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Juyoung Lee, Professor, Inha University Hospital
Other Study IDs: NAVA-Turku01
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Premature Infants; Neurally Adjusted Ventilatory Assist; Ventilator Lung; Newborn; Mechanical Ventilation
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Neurally adjusted ventilatory assist ventilation mode — This technique uses the electrical activity of the diaphragm (Edi) to control respiratory support and the NAVA level as an amplification factor that converts the Edi signal into a proportional pressure.

SUMMARY:
For the infant participating the study, ventilator settings and respiratory variables will be recorded every day and exported to a specific computer using the Servo Record Viewer version 1.0 (Maquet Critical Care AB, Getinge, Gothenburg, Sweden). Collected data gives the value for peak inspiratory pressure (PIP), expiratory tidal volume (Vt), peak Edi, minimum Edi, measured respiratory rate (RR), neural respiratory rate (nRR) and percentage of backup breaths for each minute. All the ventilator data will be inspected and compared with the event logs recorded automatically from the ventilator, which includes all the alarm notification, mode and setting changes, cables connection and disconnection data. Data during disconnection of the Edi cable, malfunction or dislocation of Edi catheter will be excluded from the analysis. The mean values during each day will be computed for each ventilatory variables. If there is a change in the ventilatory setting parameters, we will choose the one which was applied for longer duration in the 24-hour time period.

The following clinical characteristics will be collected from medical records: gestational age at birth, birth weight, gender, the time and amount of feeding, medication during the study days, desaturation events, bradycardia events, suction time and methods.

ELIGIBILITY:
Inclusion Criteria:

* babies who receiving respiratory support with neurally adjusted ventilatory assist
* babies with informed consents from their parents

Exclusion Criteria:

* babies using anesthetic agents

Ages: 0 Days to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We included preterm infants born before 36 weeks of gestation who received at least 24 hours of ventilatory support with invasive or non-invasive NAVA using a Servo-i or Servo-n ventilator (Getinge, Gothenburg, Sweden).
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
the amount of backup breaths by the ventilator | during the respiratory support using NAVA, from day 1 until the end of 36 weeks of postmenstrual age
  % time of backup/min according to babies' weight, postmenstrual age and postnatal age

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital Neonatal Intensive Care Unit, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee J, Parikka V, Lehtonen L, Soukka H. Backup ventilation during neurally adjusted ventilatory assist in preterm infants. Pediatr Pulmonol. 2021 Oct;56(10):3342-3348. doi: 10.1002/ppul.25583. Epub 2021 Jul 26. PMID 34310871